CLINICAL TRIAL: NCT00689013
Title: The Effect of Pharmacist Intervention on the Use of Zostavax in a Community Pharmacy Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); American Pharmacists Association (Other)
Responsible Party: Lindsay J. Ford, Pharm.D./Community Pharmacy Resident, University of Tennessee Community Pharmacy Residency Program
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 8750
Record Dates: First submitted 2008-05-21; First posted 2008-06-03 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Prevention & control; Pharmacists; Pharmacy; Pharmacies; Aged; Immunization; Vaccination
MeSH Terms: conditions — Herpes Zoster | interventions — College Fraternities and Sororities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Patients voluntarily presenting to community pharmacies who request receipt of the herpes zoster vaccine during the first month of observation. These patients have not been exposed to pharmacist-driven interventions utilized in this study. This group serves as the control group.
- 2 (Experimental): Patients voluntarily presenting to community pharmacies who request receipt of the herpes zoster vaccine during the second month of observation. These patients may or may not have been exposed to pharmacist-driven interventions utilized in this study. This group serves as the study/intervention group.
  Interventions: Other: Personalized letter; Other: Flyer advertisement; Other: Newspaper press release

INTERVENTIONS:
Other: Personalized letter — On Day 1 of the 2nd month, a personalized letter (addressing specific patient) was mailed to current pharmacy patients with indications for the Zostavax vaccine. Current patients were defined as those receiving at least one prescription medication from the pharmacy within 6 months. The personalized letter provided detailed information about herpes zoster infection, the vaccine for herpes zoster prevention, indications for vaccine receipt and contraindications for vaccine receipt.
  Other Names: Letter
  Arms: 2
Other: Flyer advertisement — Beginning on Day 1 of the 2nd month, flyer advertisements were distributed with all pharmacy sales. Flyer advertisements provided detailed information about herpes zoster infection, the vaccine for herpes zoster prevention, indications for vaccine receipt and contraindications for vaccine receipt.
  Other Names: Flyer
  Arms: 2
Other: Newspaper press release — During the first week of the 2nd month, local newspapers published press releases. The press release provided detailed information about herpes zoster infection, the vaccine for herpes zoster prevention, indications for vaccine receipt and contraindications for vaccine receipt.
  Other Names: Newspaper Ad
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether pharmacist-driven patient interventions can have an effect on the number of herpes zoster (Zostavax) vaccinations given in a community pharmacy setting.

DETAILED DESCRIPTION:
Several studies exist documenting the perception and satisfaction of patients receiving immunizations from pharmacists, as well as the effects of pharmacist involvement in advocating and administering vaccinations. The most well documented studies have been conducted in hospital settings. Undoubtedly, there is enormous opportunity for the community pharmacist to identify potential vaccine recipients, advocate immunization and administer said immunizations to their established patient populations. However, there is a lack of concentrated study in the implementation of immunization services in the community setting and their effects. The investigators intend to evaluate the intervention of pharmacists in an immunization program and the resulting changes in immunization rates.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 60 or older without contraindications for the herpes zoster vaccination
* patients who have already experienced one or more episodes of herpes zoster infection were considered for vaccine receipt and study inclusion secondary to CDC ACIP recommendations

Exclusion Criteria:

* Patients aged < 60 years
* Anyone who has previously received the herpes zoster vaccine
* Anyone with an allergy to neomycin, gelatin or any other component of the vaccine
* Anyone receiving a live vaccine within 4 weeks
* Anyone with a compromised or weakened immune systems such as those receiving radiation, corticosteroids, or those with HIV/AIDS, cancer in the lymph, bone or blood systems
* Pregnant women or those in close contact with a pregnant woman

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To assess the effect of a pharmacist-driven immunization campaign on the rate of Zostavax immunizations in three separate community pharmacy settings | 2 months

SECONDARY OUTCOMES:
To evaluate the relative efficacy of specific interventions on the rate of herpes zoster vaccinations | 2 months
To evaluate the perception of patients receiving the herpes zoster vaccination as to the role of pharmacists as immunizers | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay J Ford, Pharm.D., Principal Investigator — University of Tennessee Community Pharmacy Residency Program; Sarah K Frank, Pharm.D., Study Chair — University of Tennessee Community Pharmacy Residency Program; Nina H Jaber, Pharm.D., Study Chair — University of Tennessee Community Pharmacy Residency Program; Stephan L Foster, Pharm.D., Study Director — University of Tennessee Community Pharmacy Residency Program; Richard Randolph, Pharm.D., Study Chair — University of Tennessee Community Pharmacy Residency Program; Steve Lane, Pharm.D., Study Chair — University of Tennessee Community Pharmacy Residency Program; Cindy T Smith, Pharm.D., Study Chair — University of Tennessee Community Pharmacy Residency Program
Locations (3):
- United States (3):
  - Wilson Pharmacy, Johnson City, Tennessee
  - Marcrom's Pharmacy, Manchester, Tennessee
  - Reeves-Sain Drug Store, Murfreesboro, Tennessee